CLINICAL TRIAL: NCT05092243
Title: Exploit the Functional Higher Neural Connectivity and Electrophysiological Intervention of Freezing of Gait in Parkinson's Disease and Supranuclear Palsy During Different Ambulatory Complexities
Brief Title: Exploit the Functional Higher Neural Connectivity and Electrophysiological Intervention of Freezing of Gait in PD and PSP During Different Ambulatory Complexities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH110-REC3-010
Record Dates: First submitted 2021-09-29; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Transcranial Direct Current Stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Experimental): In transcranial direct current stimulation, the anodal pad was tapped over the primary motor cortex and the cathode pad was adhered of the contralateral frontal region. A constant current of 2.0 mA will be apply for up to 20 mins.
  Interventions: Device: Transcranial direct current stimulation
- sham tDCS (Sham Comparator): In transcranial direct current stimulation, the sham stimulation will be 30s stimulation with ramp up and ramp off for 10s at 2.0 mA.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — A consecutive 5-days course of tDCS will be delivered. In treatment group, true stimulation will be administrated and sham stimulation will be delivered in control group.

SUMMARY:
In the current proposal, investigators will investigate three crucial issues of FOG. Firstly, investigators will identify the possible source(s) of FOG in PD and PSP patients during unconstrained walking using a 64-channel ambulatory recorder. The investigators will explore the electric neural sources of FOG and brain connectivity. Secondarily, fMRI during motor imagery will be performed to examine the brain regions involved in the FOG patients. The investigators will merge the electrophysiological and imaging findings to detect the possible neurovascular coupling or uncoupling. Thirdly, electric intervention with transcranial direct current stimulation (tDCS) will be conducted to see whether the FOG situation can be ameliorated in PD and PSP patients. The investigators will deliver a 5-day session of tDCS to the leg motor cortex of the FOG patients to examine whether the intervention will benefit the patients in a double blind randomized design. Six assessments with different combinations of clinical scaling, gait analysis, electrophysiological investigation and fMRI examinations before and after tDCS will be conducted. Besides, there is no long-term cohort investigation of tDCS on neurodegenerative patients with FOG. The investigators will have a 3-year follow-up with a 1-month interval open-label stimulation paradigm for the patients who remained voluntarily after the termination of the initial short-term trials.

DETAILED DESCRIPTION:
The main goal of the first part of the 3-year project is to identify the source(s) of FOG with electrophysiological recording. The investigators will conduct concomitant high density Electroencephalographic and leg electromyographic recording to investigate subjects with and without FOG under unrestrained walking in the gait laboratory. The acquisitive signals from 64 montages will be decomposed first by independent component analysis (ICA) for further source localization of FOG. The event (FOG) related synchronization and desynchronization of different frequency bands of EEG will also be investigated to understand the neurophysiological implications of brain wave oscillations for the generation of FOG. In addition, the cerebello-thalamo-cortical pathway function will be assessed with magnetic paired associative stimulation in patients to probe the role of cerebellum in the pathogenesis of FOG. In the second part of the project, fMRI study will be adopted by having the subjects perform video-guided motor imagery of simple and complex walking situations. Block design paradigms will be delivered for signal acquisition. The signals will be analyzed by ICA before further processing for activation analysis. The connectivity map will beoverlaid with that of electric recording to examine the neurovascular coupling or uncoupling. In the third part of the project, investigators will deliver a 5-day session of transcranial direct current stimulation (tDCS) to the leg motor cortex of the FOG patients to examine whether the intervention will benefit the patients in a doubleblind randomized cross-over design.

ELIGIBILITY:
Inclusion Criteria:

Patients meet the diagnosis of PD or PSP based on the established consensus criteria

Exclusion Criteria:

1. Impairment of cognition that leads unable to fully cooperate with the oral commands during examinations
2. Functional III or above congestive heart failure, or cancer with distant metastasis
3. Hoehn and Yahr stage 5 in PD or PSP

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram recording before and after the tDCS session | baseline / 2 days, 2 and 4 weeks after the end of the tDCS session
  Gait recording by 64 channels EEG device. Four different frequency bands ( theta, alpha, beta, and gamma) will be investigated. Variables in gait analysis: 1.Gait initiation, 2.Level walking, 3.Gait termination.
Electromyography recording before and after the tDCS session | baseline / 2 days, 2 and 4 weeks after the end of the tDCS session
  The 4 pairs of leg EMG recording during 50 meters walking. The EMG signals will be filtered with a band pass ranging from 0.05 to 70 Hz. Variables in gait analysis: 1.Gait initiation, 2.Level walking, 3.Gait termination.
Functional magnetic resonance images examination before and after the tDCS session | baseline / 2 days after the end of the tDCS session
  fMRI scan will be performed on a 3.0T MR imager to detect the brain BOLD signal change in FOG. When fMRI was conducted, four different video tapes will be presented to the subjects：1.normal walking, 2.normal turning, 3.FOG during forward straight walking and 4.FOG during turning.

SECONDARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III before and after the tDCS session | baseline / 2 days, 2 and 4 weeks after the end of the tDCS session
  UPDRS contains four parts, the third part of which is reported in this outcome. Part III is clinician-scored monitored motor evaluation (14 questions, ranges from 0=normal to 4= Severe). The scoring of Part III varies between 0-56. The higher score indicates the worse motor function. Negative change from baseline values indicate improvement.
Change in Progressive Supranuclear Palsy Rating Scale (PSPRS) | baseline / 2 days, 2 and 4 weeks after the end of the tDCS session
  PSPRS is composed of 28 questions, divided into 6 parts: History, Mentation, Bulbar, Ocular, Limb and Gait. The scores are weighted sums of the questions in each section. Scores range from 0-100 (higher scores = more disability, lower scores = less disability). Negative change from baseline values indicate improvement.

OTHER OUTCOMES:
Change in New freezing of gait questionnaire (NFOG-Q) before and after the tDCS session | baseline / 4 weeks after the end of the tDCS session
  NFOG-Q contains three parts: in the first part, a video clip will be shown to the participants with PD and help to classify whether an individual is a freezer or non-freezer. The second and third part of the questionnaire is designed for freezers only. Par II (items 2-6, scores range between 0-19) assesses the severity of FOG according to the frequency and duration of the freezing episodes. Part III (items 7-9, scores range between 0-9) evaluates the impact of freezing on daily activities. The higher score indicates the worse freezing of gait. Negative change from baseline values indicate improvement.
Change in Tinetti's Mobility Index total score before and after the tDCS session | baseline / 4 weeks after the end of the tDCS session
  The Tinetti's Mobility Index contains two parts, Part I is Balance tests (9 questions, scores range between 0-16) and Part II is Gait tests (7 questions, scores range between 0-12). The scoring of this scale varies between 0 and 28 (< 19 high fall risk, 19-24 medium fall risk, 25-28 low fall risk). Positive change from baseline values indicate improvement.
Change inParkinson's Disease Questionnaire 39 (PDQ-39) before and after the tDCS session | baseline / 4 weeks after the end of the tDCS session
  PDQ-39 is composed of 39 questions, divided into 8 parts: mobility, activities of daily living (ADLs), emotional well-being, stigma, social support, cognition, communication and physical discomfort. It assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living. All questions range from 0 to 4 (0=never, 4=always). The scoring of this scale varies between 0-156. Negative change from baseline values indicate better quality of life rating.
Non-Motor Symptoms Questionnaire (NMSQ) | baseline / 4 weeks after the end of the tDCS session
  Non-Motor Symptoms Scale for Parkinson's Disease is composed of 30 questions, divided into 9 parts: Cardiovascular including falls, Sleep/fatigue, Mood/cognition, Perceptual problems/hallucinations, Attention/memory, Gastrointestinal tract, Urinary, Sexual function and Miscellaneous. The scoring method is frequency x severity (higher scores = more disability, lower scores = less disability). Negative change from baseline values indicate improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Chon-Haw Tsai, PHD, Principal Investigator — The chief, Department of Neurology, China Medical University Hospital
Locations (1):
- China Medical University Hospital/Neuro Depart, Taichung, Taiwan